CLINICAL TRIAL: NCT03118739
Title: Effects of Intensive Uric Acid Lowering Therapy With RDEA3170 (Verinurad) and Febuxostat in Patients With Albuminuria
Brief Title: Intensive Uric Acid Lowering With Verinurad and Febuxostat in Patients With Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5495C00007
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Hyperuricemia; Albuminuria; Type 2 Diabetes
MeSH Terms: conditions — Hyperuricemia; Albuminuria; Diabetes Mellitus, Type 2 | interventions — verinurad; Febuxostat

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, double-dummy, placebo-controlled, parallel, independent groups, repeated measures, multi-center study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Verinurad capsules/matching placebo capsules and febuxostat/matching placebo capsules with randomization code printed on each label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verinurad 9 mg+Febuxostat 80 mg (Experimental): Capsule administered orally, once daily for 24 weeks
  Interventions: Drug: Verinurad 9 mg+Febuxostat 80 mg
- Placebo (Placebo Comparator): Capsule administered orally, once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verinurad 9 mg+Febuxostat 80 mg — Capsule administered orally, once daily for 24 weeks
  Other Names: Verinurad (RDEA3170), Febuxostat(Uloric)
  Arms: Verinurad 9 mg+Febuxostat 80 mg
Drug: Placebo — Capsule administered orally, once daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this clinical research study is to evaluate signals of potential clinical benefit of the combination of Verinurad and Febuxostat in lowering concentrations of circulating uric acid and thus improving kidney or cardiovascular status of patients with hyperuricemia, albuminuria, and Type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
Evidence shows independent associations between elevated serum uric acid (sUA) and the risk of hypertension, myocardial infarction (MI), chronic kidney disease (CKD), T2DM, heart failure (HF), and metabolic syndrome, including obesity. Gout is associated with an increased risk of all-cause death, as well as cardiovascular death. The causal relationship between elevated sUA, gout, and these disease outcomes remains to be proven.

Verinurad (RDEA3170), is a novel Urate Transporter 1 (URAT1) inhibitor in Phase II development. Verinurad combined with the xanthine oxidase (XO) inhibitor febuxostat has been shown to lower sUA in patients with recurrent gout in Phase II studies by >80%. The extensive lowering of sUA delivered by the combination presents a unique opportunity to explore whether intensive urate lowering therapy can improve kidney and/or cardiac health.

This study will assess if intensive serum urate lowering therapy, more potent than ever explored before in the chronic out-patient setting, can improve chronic kidney or cardiac function in the study population.

In order to maximize the scientific value of the study and minimize the risk for systemic biases a parallel group, double blind, randomized design will be utilized.

The study will recruit patients with hyperuricemia and presenting with albuminuria.

Hyperuricemic patients are expected to benefit more from urate lowering, and albuminuria at baseline is required, as the primary objective of the study will be to assess changes in albuminuria.

Patients are also required to be diagnosed with T2DM. Patients with T2DM frequently exhibit changes in cardiac function detectable using magnetic resonance imaging (MRI) that represents an early, pre-symptomatic state of HF. By limiting recruitment to patients with T2DM and by performing MRI at baseline and 6 months of therapy, the study will deliver insights into whether or not intensive urate lowering therapy can positively affect not only chronic kidney disease, but also cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Serum Uric Acid ≥6.0 mg/dL
* eGFR ≥30 mL/min/1.73 m2
* UACR between 30 mg/g and 3500 mg/g inclusive
* Diagnosed with T2DM

Exclusion Criteria:

* Treated with any drug for hyperuricemia in the 6 months preceding randomization.Drugs for hyperuricemia include all XO inhibitors (allopurinol, febuxostat and topiroxostat) and URAT1 inhibitors (lesinurad, verinurad, probenecid, and benzbromarone)
* Prior history of gout, unless prophylaxis therapy isn't required
* Patients who are pregnant, lactating, or planning to become pregnant
* Patients unsuitable or unable to undergo MRI assessment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Site, Canyon Country, California
  - Research Site, Chula Vista, California
  - Research Site, Corona, California
  - Research Site, Escondido, California
  - Research Site, Lakewood, California
  - Research Site, Lincoln, California
  - Research Site, Los Angeles, California
  - Research Site, North Hollywood, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, Houston, Texas
  - Research Site, Pearland, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Webster, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will likely not be shared with external collaborators/researchers as this data is planned to be used only for internal decision-making

REFERENCES:
- [Derived] Heerspink HJL, Stack AG, Terkeltaub R, Greene TA, Inker LA, Bjursell M, Perl S, Rikte T, Erlandsson F, Perkovic V. Rationale, design, demographics and baseline characteristics of the randomized, controlled, Phase 2b SAPPHIRE study of verinurad plus allopurinol in patients with chronic kidney disease and hyperuricaemia. Nephrol Dial Transplant. 2022 Jul 26;37(8):1461-1471. doi: 10.1093/ndt/gfab237. PMID 34383954
- [Derived] Stack AG, Dronamraju N, Parkinson J, Johansson S, Johnsson E, Erlandsson F, Terkeltaub R. Effect of Intensive Urate Lowering With Combined Verinurad and Febuxostat on Albuminuria in Patients With Type 2 Diabetes: A Randomized Trial. Am J Kidney Dis. 2021 Apr;77(4):481-489. doi: 10.1053/j.ajkd.2020.09.009. Epub 2020 Oct 29. PMID 33130235
- See also: Redacted Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00007&attachmentIdentifier=7ba9d99a-a3d8-4550-9897-42c1821775ff&fileName=d5495c00007_csp_Redacted.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00007&attachmentIdentifier=fe54e85c-c086-4dca-89de-900472089931&fileName=d5495c00007_sap_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 19 clinical research centers in the United States of America. First subject enrolled (First subject first visit/first consent signed date): 18 May 2017. Last subject last visit: 13 August 2018.
Pre-assignment Details: Patients were screened at Visit 1. Within 1 week, eligible patients collected 3 morning void samples on consecutive days for proteinuria measurements. Patients with acceptable results were scheduled for Visit 2. Prior to randomization and before or on the day of Visit 2, patients underwent MRI. V2 occurred no later than 6 weeks after V1.
Period: Overall Study
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Started | 32 | 28
Completed 12 Weeks of Treatment | 26 | 25
Completed 24 Weeks of Treatment | 24 | 25
Completed | 25 | 24
Not Completed | 7 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Categorical [Count of Participants; unit: Participants] — Age at Randomization
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 16 | 17 | 33
    >=65 years | 16 | 11 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening
  Years | 62.0 (9.51) | 60.9 (12.15) | 61.5 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 22 | 20 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 18
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 5 | 11
  White | 22 | 15 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Weight [Mean (Standard Deviation); unit: kg] | 93.72 (20.243) | 96.76 (19.561) | 95.14 (19.818)
Height [Mean (Standard Deviation); unit: cm] | 170.57 (10.662) | 170.75 (9.117) | 170.65 (9.888)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 32.00 (5.082) | 32.95 (4.699) | 32.44 (4.889)
estimated glomerular filtration rate (eGFR) [Count of Participants; unit: Participants]
  eGFR<30 | 2 | 1 | 3
  eGFR >=30 to <60 | 16 | 9 | 25
  eGFR >=60 to <90 | 9 | 12 | 21
  eGFR >=90 | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Urinary Albumin to Creatinine Ratio (UACR)
Description: LS Mean Percentage Change (95% CI) from Baseline in UACR
Time Frame: From Baseline to 12 Weeks of Treatment
Population: Number analyzed at 12 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Precent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Precent change | -48.65 [-64.807 to -25.089] | -15.31 [-43.244 to 26.370]
Statistical Analysis 1: Comparison: Verinurad 9 mg+Febuxostat 80 mg vs Placebo; Test type: Superiority; Mean % Change from Baseline = -39.37, 90% CI 2-sided [-61.785 to -3.814]

2. Secondary Outcome: sUA
Description: LS Mean Percentage Change (95% CI) from Baseline in sUA
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Percent change
  12 weeks: number analyzed (Participants) | 30 | 26
  12 weeks | -56.81 [-63.879 to -48.350] | 6.86 [-11.800 to 29.471]
  24 weeks: number analyzed (Participants) | 27 | 24
  24 weeks | -61.93 [-68.274 to -54.319] | 4.73 [-13.795 to 27.239]

3. Secondary Outcome: eGFR
Description: LS Mean Percentage Change (95% CI) from Baseline in eGFR
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Percent change
  12 weeks: number analyzed (Participants) | 30 | 26
  12 weeks | 1.25 [-6.520 to 9.674] | -4.40 [-12.258 to 4.154]
  24 weeks: number analyzed (Participants) | 27 | 24
  24 weeks | -1.73 [-9.446 to 6.648] | 0.55 [-7.854 to 9.712]

4. Secondary Outcome: Serum Creatinine
Description: LS Mean Percentage Change (95% CI) from Baseline in Serum Creatinine
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Percent change
  12 weeks: number analyzed (Participants) | 30 | 26
  12 weeks | -0.60 [-6.946 to 6.188] | 3.44 [-3.636 to 11.025]
  24 weeks: number analyzed (Participants) | 27 | 24
  24 weeks | 1.93 [-4.743 to 9.078] | 0.02 [-6.945 to 7.504]

5. Secondary Outcome: Serum Cystatin C
Description: LS Mean Percentage Change (95% CI) from Baseline in Serum Cystatin C
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Percent change
  12 weeks: number analyzed (Participants) | 30 | 26
  12 weeks | 3.252 [-1.3402 to 8.0581] | 0.114 [-4.6520 to 5.1187]
  24 weeks: number analyzed (Participants) | 27 | 24
  24 weeks | 5.412 [0.5212 to 10.5418] | 3.951 [-1.1612 to 9.3279]

6. Secondary Outcome: Serum High Sensitivity C-reactive Protein
Description: LS Mean Percentage Change (95% CI) from Baseline in Serum High Sensitivity C-reactive Protein
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Percent change
  12 weeks: number analyzed (Participants) | 30 | 26
  12 weeks | 35.863 [4.5883 to 76.4884] | 11.665 [-15.6408 to 47.8091]
  24 weeks: number analyzed (Participants) | 27 | 24
  24 weeks | -8.002 [-29.9761 to 20.8680] | 9.793 [-17.8132 to 46.6716]

7. Secondary Outcome: Clinical Assessments
Description: Change from Baseline in Diastolic and Systolic Blood Pressure
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mm/Hg
  Diastolic BP, mmHg Baseline | 74.7 (9.83) | 77.8 (11.91)
  Diastolic BP, mmHg 12 weeks (Change from baseline): number analyzed (Participants) | 29 | 25
  Diastolic BP, mmHg 12 weeks (Change from baseline) | 1.6 (11.02) | -0.2 (9.51)
  Diastolic BP, mmHg 24 weeks (Change from baseline): number analyzed (Participants) | 28 | 25
  Diastolic BP, mmHg 24 weeks (Change from baseline) | 2.0 (8.53) | 1.7 (12.05)
  Systolic BP, mmHg Baseline | 136.4 (15.13) | 138.5 (16.34)
  Systolic BP, mmHg 12 weeks (Change from baseline): number analyzed (Participants) | 29 | 25
  Systolic BP, mmHg 12 weeks (Change from baseline) | -0.8 (19.00) | -3.2 (15.48)
  Systolic BP, mmHg 24 weeks (Change from baseline): number analyzed (Participants) | 28 | 25
  Systolic BP, mmHg 24 weeks (Change from baseline) | 0.4 (9.75) | -0.6 (17.78)

8. Secondary Outcome: MRI Variables - LV Mass/End-diastolic Volume
Description: Change from Baseline in MRI Variables at Week 24 (CFB = Change from Baseline)
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: g/mL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
g/mL | 0.049 (0.1445) | 0.053 (0.1202)

9. Other Pre Specified Outcome: Flow Mediated Dilatation (Reactive Hyperemia)
Description: LS Mean Change (95% CI) from Baseline in Flow Mediated Dilatation. The flow mediated dilatation metric is obtained using a device from Cordex, and a proprietary algorithm.
  This metric represents the volume difference between a baseline arterial compliance curve and hyperemia arterial compliance curve in the positive transmural pressure region. This metric has a direct relationship to a subject's cardiovascular condition. Output range is 0-150. A higher score is indicative of a better flow mediated dilatation.
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Units on a scale
  12 weeks Change from Baseline: number analyzed (Participants) | 22 | 23
  12 weeks Change from Baseline | 0.8 [-10.59 to 12.24] | -5.9 [-17.04 to 5.29]
  24 weeks Change from Baseline: number analyzed (Participants) | 19 | 19
  24 weeks Change from Baseline | 0.5 [-9.44 to 10.47] | -5.5 [-15.47 to 4.44]

10. Other Pre Specified Outcome: Urinalysis
Description: Changes in Urinalysis (CFB = Change from Baseline)
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/dL
  Baseline Protein, mg/dL: number analyzed (Participants) | 28 | 25
  Baseline Protein, mg/dL | 72.01 (99.767) | 65.74 (78.686)
  Protein, mg/dL 12 weeks (CFB): number analyzed (Participants) | 25 | 23
  Protein, mg/dL 12 weeks (CFB) | -11.40 (65.896) | -4.07 (71.047)
  Protein, mg/dL 24 weeks (CFB): number analyzed (Participants) | 23 | 22
  Protein, mg/dL 24 weeks (CFB) | -16.73 (101.052) | 11.40 (76.645)
  Baseline Urine Albumin, mg/dL | 38.0907 (55.62178) | 35.8905 (47.17446)
  Urine Albumin, mg/dL 12 weeks (CFB): number analyzed (Participants) | 29 | 26
  Urine Albumin, mg/dL 12 weeks (CFB) | -9.4766 (35.73442) | -0.3019 (45.81688)
  Urine Albumin, mg/dL 24 weeks (CFB): number analyzed (Participants) | 27 | 24
  Urine Albumin, mg/dL 24 weeks (CFB) | -6.9482 (50.66844) | 11.6049 (53.13042)
  Baseline Urine Creatinine, mg/dL | 96.52 (51.570) | 86.25 (46.189)
  Urine Creatinine, mg/dL 12 weeks (CFB): number analyzed (Participants) | 29 | 26
  Urine Creatinine, mg/dL 12 weeks (CFB) | 5.06 (53.378) | 12.95 (34.987)
  Urine Creatinine, mg/dL 24 weeks (CFB): number analyzed (Participants) | 27 | 24
  Urine Creatinine, mg/dL 24 weeks (CFB) | 7.58 (55.930) | 8.53 (36.430)
  Baseline Urine Urate, mg/dL: number analyzed (Participants) | 28 | 25
  Baseline Urine Urate, mg/dL | 28.354 (12.0591) | 23.960 (10.6862)
  Urine Urate, mg/dL 12 weeks (CFB): number analyzed (Participants) | 25 | 23
  Urine Urate, mg/dL 12 weeks (CFB) | -13.394 (13.2757) | 3.560 (12.3875)
  Urine Urate, mg/dL 24 weeks (CFB): number analyzed (Participants) | 23 | 22
  Urine Urate, mg/dL 24 weeks (CFB) | -10.732 (16.4720) | 2.294 (9.3407)

11. Other Pre Specified Outcome: Clinical Chemistry Values
Description: Changes in Clinical Chemistry Values (CFB = Change for Baseline)
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
pmol/L
  Baseline Aldosterone, pmol/L: number analyzed (Participants) | 31 | 28
  Baseline Aldosterone, pmol/L | 134.58 (126.126) | 95.11 (72.640)
  Aldosterone, pmol/L 12 weeks (CFB): number analyzed (Participants) | 27 | 26
  Aldosterone, pmol/L 12 weeks (CFB) | 1.12 (118.622) | 14.72 (72.485)
  Aldosterone, pmol/L 24 weeks (CFB): number analyzed (Participants) | 24 | 24
  Aldosterone, pmol/L 24 weeks (CFB) | 9.14 (102.932) | 38.14 (90.007)
  Baseline NT-proBNP, pmol/L: number analyzed (Participants) | 29 | 27
  Baseline NT-proBNP, pmol/L | 23.230 (22.6864) | 15.866 (28.2147)
  NT-proBNP, pmol/L 12 weeks (CFB): number analyzed (Participants) | 25 | 25
  NT-proBNP, pmol/L 12 weeks (CFB) | 4.621 (31.1027) | 1.556 (10.0140)
  NT-proBNP, pmol/L 24 weeks (CFB): number analyzed (Participants) | 24 | 21
  NT-proBNP, pmol/L 24 weeks (CFB) | 6.267 (19.0367) | 15.866 (46.4392)

12. Primary Outcome: Urinary Albumin to Creatinine Ratio (UACR) Compared to Placebo
Description: LS Mean Percentage Change (90% CI) from Baseline in UACR Compared to Placebo
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (90% Confidence Interval); unit: Precent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Precent change | -49.26 [-68.206 to -19.009] | NA [NA to NA] — The primary endpoint is a comparison

13. Secondary Outcome: MRI Variables - Kidney Cortex T2 Star - BOLD MRI
Description: Change from Baseline in MRI Variables at Week 24 (CFB = Change from Baseline)
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
ms | -1.46 (6.511) | -1.67 (6.440)

14. Secondary Outcome: MRI Variables - LV End-diastolic Volume, LV End-systolic Volume, LV Stroke Volume
Description: Change from Baseline in MRI Variables at Week 24 (CFB = Change from Baseline)
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mL
  LV End-diastolic Volume (mL) (CFB): number analyzed (Participants) | 18 | 15
  LV End-diastolic Volume (mL) (CFB) | -5.39 (27.458) | -4.93 (20.665)
  LV End-systolic Volume (mL) (CFB): number analyzed (Participants) | 18 | 15
  LV End-systolic Volume (mL) (CFB) | 1.33 (14.106) | -2.48 (10.703)
  LV Stroke Volume (mL) (CFB): number analyzed (Participants) | 18 | 15
  LV Stroke Volume (mL) (CFB) | -6.73 (15.923) | -2.44 (12.458)

15. Secondary Outcome: MRI Variables - LV Ejection Fraction, Circumferential Strain, Longitudinal Strain, Radial Strain
Description: Change from baseline in MRI Variables at Week 24 (CFB = Change from Baseline)
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: % (change in percentage from baseline)
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
% (change in percentage from baseline)
  LV Ejection Fraction (%) (CFB): number analyzed (Participants) | 18 | 15
  LV Ejection Fraction (%) (CFB) | -2.08 (3.761) | 0.59 (3.374)
  Circumferential Strain (%) (CFB): number analyzed (Participants) | 18 | 15
  Circumferential Strain (%) (CFB) | -0.25 (2.321) | -0.07 (2.192)
  Longitudinal Strain (%) (CFB): number analyzed (Participants) | 19 | 15
  Longitudinal Strain (%) (CFB) | 0.29 (1.949) | 0.53 (1.729)
  Radial Strain (%) (CFB): number analyzed (Participants) | 18 | 15
  Radial Strain (%) (CFB) | -2.29 (7.136) | 1.44 (8.109)

16. Secondary Outcome: MRI Variables - Diastolic Circumferential Strain Rate, Longitudinal Strain Rate, Radial Strain Rate and Systolic Circumferential Strain Rate, Longitudinal Strain Rate, Radial Strain Rate
Description: Change from Baseline in MRI Variables at Week 24 (CFB = Change from Baseline)
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
s^-1
  Diastolic Circumferential Strain Rate (s^-1) (CFB): number analyzed (Participants) | 18 | 15
  Diastolic Circumferential Strain Rate (s^-1) (CFB) | -0.0496 (0.13769) | -0.0384 (0.13791)
  Diastolic Longitudinal Strain Rate (s^-1) (CFB): number analyzed (Participants) | 19 | 15
  Diastolic Longitudinal Strain Rate (s^-1) (CFB) | -0.0043 (0.10629) | -0.0300 (0.16940)
  Diastolic Radial Strain Rate (s^-1) (CFB): number analyzed (Participants) | 18 | 15
  Diastolic Radial Strain Rate (s^-1) (CFB) | 0.2348 (0.43676) | 0.0201 (0.72927)
  Systolic Circumferential Strain Rate (s^-1) (CFB): number analyzed (Participants) | 18 | 15
  Systolic Circumferential Strain Rate (s^-1) (CFB) | 0.0115 (0.11314) | -0.0743 (0.11616)
  Systolic Longitudinal Strain Rate (s^-1) (CFB): number analyzed (Participants) | 19 | 15
  Systolic Longitudinal Strain Rate (s^-1) (CFB) | 0.0285 (0.08436) | -0.0021 (0.08052)
  Systolic Radial Strain Rate (s^-1) (CFB): number analyzed (Participants) | 18 | 15
  Systolic Radial Strain Rate (s^-1) (CFB) | -0.1917 (0.31833) | 0.2516 (0.38049)

17. Secondary Outcome: MRI Variables - LV Mass
Description: Change from Baseline in MRI Variables at Week 24 (CFB = Change from Baseline)
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
g | 1.80 (7.532) | 2.63 (9.994)

18. Other Pre Specified Outcome: Urinalysis
Description: Changes in Urinalysis (CFB = Change from Baseline)
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/g
  Baseline Protein/Creatinine, mg/g: number analyzed (Participants) | 27 | 25
  Baseline Protein/Creatinine, mg/g | 945.56 (1457.714) | 828.52 (987.671)
  Protein/Creatinine, mg/g 12 weeks (CFB): number analyzed (Participants) | 22 | 23
  Protein/Creatinine, mg/g 12 weeks (CFB) | -185.33 (366.340) | -155.44 (584.772)
  Protein/Creatinine, mg/g 24 weeks (CFB): number analyzed (Participants) | 21 | 19
  Protein/Creatinine, mg/g 24 weeks (CFB) | -98.60 (397.778) | 177.11 (1387.627)

19. Other Pre Specified Outcome: Clinical Chemistry Values
Description: Changes in Clinical Chemistry Values (CFB = Change for Baseline)
Time Frame: From Baseline to 12 Weeks and 24 Weeks of Treatment
Population: Number analyzed at 12 and 24 weeks was less than the overall number analyzed due to missing observations
Measure: Mean (Standard Deviation); unit: % hemoglobin bound to glucose
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
% hemoglobin bound to glucose
  Baseline Hemoglobin A1C/Hemoglobin, %: number analyzed (Participants) | 32 | 27
  Baseline Hemoglobin A1C/Hemoglobin, % | 8.14 (1.913) | 8.28 (2.025)
  Hemoglobin A1C/Hemoglobin, % 12 weeks (CFB): number analyzed (Participants) | 30 | 25
  Hemoglobin A1C/Hemoglobin, % 12 weeks (CFB) | 0.20 (1.399) | 0.13 (1.159)
  Hemoglobin A1C/Hemoglobin, % 24 weeks (CFB): number analyzed (Participants) | 27 | 21
  Hemoglobin A1C/Hemoglobin, % 24 weeks (CFB) | -0.14 (0.884) | 0.22 (1.863)

20. Other Pre Specified Outcome: Baseline eGFR
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mL/min/1.73m2 | 59.2 (25.25) | 68.1 (23.15)

21. Other Pre Specified Outcome: Baseline UACR
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/g | 459.05 (824.731) | 411.55 (547.816)

22. Other Pre Specified Outcome: Baseline Serum Uric Acid (sUA)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/dL | 7.51 (1.558) | 7.02 (0.813)

23. Other Pre Specified Outcome: Baseline Serum Creatinine
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/dL | 1.40 (0.595) | 1.19 (0.362)

24. Other Pre Specified Outcome: Baseline Serum Cystatin-C
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/L | 1.579 (0.5274) | 1.313 (0.3532)

25. Other Pre Specified Outcome: Baseline Serum High-sensitivity C-reactive Protein
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
mg/dL | 0.410 (0.3670) | 0.358 (0.2506)

26. Other Pre Specified Outcome: Baseline MRI Variables - Kidney Cortex T2 Star
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 27
ms | 81.13 (12.995) | 82.31 (11.625)

27. Other Pre Specified Outcome: Baseline MRI Variables - LV End-diastolic Volume
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
mL | 161.47 (37.766) | 161.50 (32.639)

28. Other Pre Specified Outcome: Baseline MRI Variables - LV Ejection Fraction
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: % (percentage of LV volume)
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
% (percentage of LV volume) | 59.77 (7.869) | 60.19 (6.134)

29. Other Pre Specified Outcome: Baseline MRI Variables - LV End-systolic Volume
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
mL | 66.43 (26.089) | 64.63 (17.977)

30. Other Pre Specified Outcome: Baseline MRI Variables - Circumferential Strain
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: % (change in percentage in LV dimension)
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
% (change in percentage in LV dimension) | -14.10 (3.925) | -15.37 (2.901)

31. Other Pre Specified Outcome: Baseline MRI Variables - Diastolic Circumferential Strain Rate
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
s^-1 | 0.6371 (0.24946) | 0.7588 (0.21276)

32. Other Pre Specified Outcome: Baseline MRI Variables - Diastolic Longitudinal Strain Rate
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
s^-1 | 0.4833 (0.21090) | 0.5258 (0.16476)

33. Other Pre Specified Outcome: Baseline MRI Variables - Diastolic Radial Strain Rate
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
s^-1 | -2.3143 (1.08926) | -2.7591 (1.05712)

34. Other Pre Specified Outcome: Baseline MRI Variables - Longitudinal Strain
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: % (change in percentage in LV dimension)
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
% (change in percentage in LV dimension) | -12.07 (3.779) | -12.21 (3.102)

35. Other Pre Specified Outcome: Baseline MRI Variables - Radial Strain
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: % (change in percentage in LV dimension)
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
% (change in percentage in LV dimension) | 43.47 (15.943) | 46.45 (12.743)

36. Other Pre Specified Outcome: Baseline MRI Variables - Systolic Circumferential Strain Rate
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
s^-1 | -0.7673 (0.19408) | -0.7797 (0.12776)

37. Other Pre Specified Outcome: Baseline MRI Variables - Systolic Longitudinal Strain Rate
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
s^-1 | -0.6278 (0.16784) | -0.6552 (0.12734)

38. Other Pre Specified Outcome: Baseline MRI Variables - Systolic Radial Strain Rate
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: s^-1
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
s^-1 | 2.1059 (0.66890) | 2.1220 (0.58484)

39. Other Pre Specified Outcome: Baseline MRI Variables - LV Mass
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
g | 110.27 (26.229) | 110.82 (28.487)

40. Other Pre Specified Outcome: Baseline MRI Variables - LV Mass/End-diastolic Volume
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: g/mL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
g/mL | 0.696 (0.1437) | 0.687 (0.1163)

41. Other Pre Specified Outcome: Baseline MRI Variables - LV Stroke Volume
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with MRI (exam not completed)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 26
mL | 95.05 (19.327) | 96.86 (21.286)

42. Other Pre Specified Outcome: Baseline Flow Mediated Dilatation (Reactive Hyperemia)
Description: Baseline in Flow Mediated Dilatation. The flow mediated dilatation metric is obtained using a device from Cordex, and a proprietary algorithm.
  This metric represents the volume difference between a baseline arterial compliance curve and hyperemia arterial compliance curve in the positive transmural pressure region. This metric has a direct relationship to a subject's cardiovascular condition. Output range is 0-150. A higher score is indicative of a better flow mediated dilatation.
Time Frame: Baseline
Population: Total number differs from Study totals due to subject non compliance with exam (exam not completed)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 29 | 26
Units on a scale | 60.4 (28.76) | 60.6 (30.90)

43. Primary Outcome: Urinary Albumin to Creatinine Ratio (UACR)
Description: LS Mean Percentage Change (95% CI) from Baseline in UACR
Time Frame: From Baseline to 24 Weeks of Treatment
Population: Number analyzed at 24 weeks was less than the overall number analyzed due to missing observations
Measure: Least Squares Mean (95% Confidence Interval); unit: Precent change
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
Number analyzed (Participants) | 32 | 28
Precent change | -38.40 [-58.051 to -9.535] | 21.40 [-18.948 to 81.829]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of signature of informed consent (Screening Visit) throughout the treatment period and including the follow-up period (Day 190).
Description: AEs were spontaneously reported by the patient or reported in response to an open question from the study site staff.
Arm/Group | Verinurad 9 mg+Febuxostat 80 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/32 | 3/28
Other Adverse Events (participants affected / at risk) | 9/32 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verinurad 9 mg+Febuxostat 80 mg (N=32) | Placebo (N=28)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Troponin I Increased (Investigations) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Wound Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verinurad 9 mg+Febuxostat 80 mg (N=32) | Placebo (N=28)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The treatment code was broken for 3 patients.The effect of verinurad/febuxostat on sUA was underestimated as drug was administered after collection of blood samples.3 patients treated with verinurad/febuxostat had no detectable drug in PK samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03118739/Prot_SAP_000.pdf